CLINICAL TRIAL: NCT05470010
Title: The SEAMLESS Study: A Pragmatic Multi-Site Randomized Waitlist-Controlled Trial of a Smartphone App-Based Mindfulness Intervention for French and English Speaker Cancer Survivors
Brief Title: Smartphone App-Based Mindfulness Intervention for French and English Speaker Cancer Survivors
Acronym: SEAMLESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SC28
Record Dates: First submitted 2022-05-19; First posted 2022-07-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Psychological
Keywords: Cancer survivors; Smartphone app; Mindfulness
MeSH Terms: conditions — Neoplasms | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Mindfulness (Experimental): A 4 week smartphone app-based mindfulness intervention program with in-app activities for 20-30 minutes everyday, with a minimum of 4 days of activity in a week.
  Interventions: Behavioral: Mindfulness
- Control Mindfulness (Other): No intervention and usual care for 4 weeks, after which there will be assessments immediately post-waiting and at 3 months post-baseline. After this, participants will get the same 4 week smartphone app-based mindfulness intervention program.
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — A psychological behavioral intervention that trains participants in mindfulness techniques, which involves achieving a moment-to-moment non-judgmental awareness of their internal psychosocial-emotional state through meditation and gentle mindful movements.

SUMMARY:
There is a need to develop, evaluate, and disseminate self-directed, easily accessible, safe, affordable, and effective psychosocial interventions to people living with cancer (PLWC) post-treatment. Smartphone app-based health interventions are an innovative way to deliver psychosocial cancer-care. The Mindfulness-Based Cancer Survivorship (MBCS) Journey app is a mobile app format of the Mindfulness-based Cancer Recovery program. In the SEAMLESS Study, the investigators aim to evaluate the MBCS Journey app (a 4 week mind-body intervention) in cancer survivors post-treatment. This is a randomized wait-list controlled trial. Participants will either be assigned into the immediate group (will receive intervention immediately after enrollment) or the waitlist group (wait for 3 months before receiving the intervention).

DETAILED DESCRIPTION:
BACKGROUND: Cancer patients who are transitioning into the survivorship phase after completing their final treatments often have unmet needs that are different than those faced during the diagnosing phase or treatment phase of their journey. PLWC tend to experience late and long-term effects such as pain, fatigue, and distress. They can also experience psychosocial stressors such as anxiety, depression, uncertainty about the future, and the fear of cancer reoccurrence, which can negatively impact their mental health.

Cancer survivors are often unable to receive the face-to-face care they need due to barriers such as compromised immunity, treatment-related side effects, scheduling conflicts, and geography. Having a smartphone app-based mind-body intervention can help patients overcome several of these barriers since they are able to participate in at their own convenience in the comfort of their own home without the burden of travelling to and scheduling these classes.

INTERVENTION DESIGN: The AM smartphone app (where MBCS Journey can be found) supports personalized mindfulness practices through lessons and personalized guided-meditation playlists. The AM app is able to interpret its users' emotional state e.g. angry, elated. from a user-inputted digital emotion-mapping board; and heart-rate data through algorithms that analyze facial bio-signals. The SEAMLESS study aims to evaluate AM's effectiveness for reducing stress (primary outcome), anxiety, depression, fatigue, and overall physical functioning and quality of life (secondary outcome) as well as determining the mechanisms of action. In addition, there are two exploratory objectives: 1) to explore the sex, and gender-based differences in significant outcomes as well as subgroup effects by cancer stage, type, ethnicity, and age and 2) explore the correlation between self-reported stress reduction and app usage and the correlation between stress ratings and psycho-biometric data collected within the app. Outcomes will be assessed using validated Calgary Symptoms of Stress Inventory (for stress), the PROMIS measure (for anxiety, depression, fatigue, and overall physical functioning), and the European Organization for Research and Treatment of Cancer quality of life questionnaire (for quality of life). Assessments will occur at 1) baseline, 2) post-intervention, 3) 3 month after baseline follow-up, and 4) 6 month post-intervention follow-up.

SIGNIFICANCE: In today's digital world, there are many app-based interventions for patients but cancer-care providers are uncertain about their efficacy. Our study will provide rigorously evaluated efficacy data for a smartphone app-based mind-body intervention for cancer survivors, which if helpful, could be made easily available for psychosocial care at cancer centers worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years
* Diagnosed with any type of cancer (stages I-IV)
* Completed primary treatment (i.e. surgery, chemotherapy, radiation therapy) at least 2 weeks (14days) prior. Note: ongoing maintenance therapy, hormone-blocking therapies, intermittent bone-modifying agents, herceptin and targeted therapy with trastuzumab are not exclusionary.
* Have access to a smartphone with data or wifi connection.
* Willing to devote 20-30 mins of time to mindfulness practices daily during the 4-week intervention period.
* Participant consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each participant must sign a consent form (e-consent) prior to enrollment in the study to document their willingness to participate.
* Participant is able (i.e. sufficiently fluent) and willing to complete the MBCS Journey and outcome measures in either English or French. The baseline assessment must be completed within required timelines, prior to randomization.
* In accordance with CCTG policy, protocol intervention is intended to begin within 7 calendar days of patient randomization.
* Participants must be willing to complete the MBCS Journey and complete the follow-up questionnaires

Exclusion Criteria:

* Major communication difficulties at the time of recruitment, as assessed by the research team (e.g. severe hearing impairment or cognitive impairment (score of ≤ 6; as assessed by the centre CRA using the three questions from the Brief Screen for Cognitive Impairment (BSCI)) listed in the screening CRF, which could interfere with completing the intervention and/or the questionnaires (i.e. inability to read or write)
* Suffering from untreated Major Depressive Disorder or other psychiatric disorders that would interfere with participation. (Note: Participants will be referred for treatment and invited to call back once in remission).
* Previous experience practicing in-person or app-based mindfulness once a week or more within the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Calgary Symptoms of Stress Inventory (C-SOSI) | 3 months
  This is a 56 item scale. Each item is rated on a 5-point Likert scale (1-5). A higher score indicates higher levels of stress.

SECONDARY OUTCOMES:
Patient Reported Outcome Measurement Information System (PROMIS) - Anxiety | 3 months
  Short form (4 items). A higher score indicates higher levels of anxiety.
Patient Reported Outcome Measurement Information System (PROMIS) - Depression | 3 months
  Short form (4 items). A higher score indicates higher levels of depression.
Patient Reported Outcome Measurement Information System (PROMIS) - Fatigue | 3 months
  Short form (4 items). A higher score indicates higher levels of fatigue.
Patient Reported Outcome Measurement Information System (PROMIS) - Physical Function | 3 months
  PROMIS - Cancer Bank v1.1 - Physical Function. This questionnaire has 45 items, each rated on a 5-point Likert scale. A higher score indicates better physical functioning.
Quality of Life - European Organization for Research and Treatment of Cancer quality of life | 3 months
  European Organization for Research and Treatment of Cancer quality of life - EORTC QLQ C-30. The two items measuring quality of life were used. Each item is rated on a 7-point Likert scale (1-7).
App-based User Data - Perceived Stress | 3 months
  Perceived stress will be measured using a stress slider within the app.
App-based User Data - Mood | 3 months
  Mood will be measured using a mood board.
App-based User Data - Objective Stress | 3 months
  Biometric imaging will be used to measure heart rate and blood flow which combined will predict the participant's "objective stress".

CONTACTS AND LOCATIONS:
Overall Officials: Linda E Carlson, Study Chair — University of Calgary
Locations (7):
- Canada (7):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - BCCA - Kelowna, Kelowna, British Columbia
  - BCCA - Prince George, Prince George, British Columbia
  - BCCA - Victoria, Victoria, British Columbia
  - Western Manitoba Cancer Centre, Brandon, Manitoba
  - Horizon Health Network, Fredericton, New Brunswick
  - Kingston Health Sciences Centre, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No